CLINICAL TRIAL: NCT06432192
Title: ApoDiag: A Prospective, Monocentric Clinical Study for the Validation of in Vitro Diagnostic Tests Developed by Firalis
Brief Title: A Prospective, Monocentric Clinical Study for the Validation of in Vitro Diagnostic Tests Developed by Firalis
Acronym: ApoDiag
Status: Completed | Type: Observational
Sponsor: Firalis SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A02120-45
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-09

CONDITIONS: Genetic Health Risks
Keywords: Polygenic risk; APOE, Apolipoprotein; Neurodegenerative disorders; Dementia; Alzheimer disease; Genetic risks
MeSH Terms: conditions — Neurodegenerative Diseases; Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- APOE E: The cohort will be genotyped to determine the phenotype of the APOE allele
  Interventions: Diagnostic Test: APO-Easy

INTERVENTIONS:
Diagnostic Test: APO-Easy — Testing for the APOE genotype using the APO-Easy Genotyping test

SUMMARY:
Firalis SA and its affiliate Amoneta Diagnostics SAS are developing novel in-vitro-diagnostic (IVD) tests for diverse diagnostic applications for major human diseases, including cardiovascular, and neurodegenerative disorders. These tests detect several gene mutations related to the above-mentioned pathologies. The development of IVD tools requires the evaluation of analytical parameters including biomarker stability.

The present specific study therefore aims to collect whole blood samples in PAXgene DNA tubes to complete the analytical validation of IVD tools and the evaluation of the stability of the DNA in PAXgene DNA tubes and the reagents in the IVD tools.

ELIGIBILITY:
Inclusion Criteria:

* Donors who sign the informed consent forms for sample collection and for genotyping.
* Adults, both genders, aged 18-85 years.
* Not under any administrative or legal supervision

Exclusion Criteria:

* Anyone who did not sign the Informed Consent form.
* Subjects aged below 18 years and older than 85 years are excluded.
* Pregnant, parturient and nursing women are excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy donors
Sampling Method: Non-Probability Sample
Enrollment: 1474 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
APOE Genotype | Baseline
  Blood samples will be collected to establish the feasibility of detecting several gene mutations associated with the risk of Alzheimer's disease/ Cardiovascular disorder and validation of analytical parameters

SECONDARY OUTCOMES:
Specimen stability | Baseline, 24hrs, 5 days, 28 days, 3 months, 12 months, 24 months
  Blood samples will be collected to establish the stability of PAXgene DNA samples at different timepoints after storage at -20° and -80°C.

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Firat, MD PhD, Study Director — Firalis SA; Lucas Pham-Van, PhD, Study Chair — Firalis SA; Joanna Michel, Study Chair — Firalis SA; Sthepanie Boutillier, PhD, Study Director — Firalis SA
Locations (2):
- France (2):
  - EFS GEST, Nancy
  - EFS GEST, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided